CLINICAL TRIAL: NCT04283383
Title: Effectiveness of a Primary Care Clinical Ultrasound Classroom for Family Physicians as a Formative Intervention System, a Cuasi Experimental Trial. Study Protocol
Brief Title: Effectiveness of a Primary Care Clinical Ultrasound Classroom
Acronym: AECAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GRS 1824 B 18
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: ULTRASONOGRAPHY; PRIMARY CARE

STUDY DESIGN:
Intervention Model Description: quasi-experimental study,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention training (Experimental): A structured training process oriented to the clinical practice of the family physician, Primary Care Clinical Ultrasound Classroom (AECAP) will be carried out, and the improvement of knowledge and skills will be evaluated, as well as the improvement of quality of care based on clinical indicators.
  Interventions: Other: Primary Care Clinical Ultrasound Classroom (AECAP)
- control (No Intervention)

INTERVENTIONS:
Other: Primary Care Clinical Ultrasound Classroom (AECAP) — A structured training process oriented to the clinical practice of the family physician, Primary Care Clinical Ultrasound Classroom (AECAP) will be carried out,
  Arms: Intervention training

SUMMARY:
Introduction: Clinical ultrasound is a technique that increases diagnostic capacity and facilitates clinical decision making. The objective is to develop and validate an ultrasound training methodology oriented to the clinical practice of the family doctor.

Methods: quasi-experimental study, with before / after design, with a control group and one year of follow-up. 20 family doctors working in primary care Health Centers and with a list of patients over 800 will be included and a control group of similar characteristics will be selected, in terms of age, gender and patient list. A structured training process oriented to the clinical practice of the family physician, Primary Care Clinical Ultrasound Classroom (AECAP) will be carried out, and the improvement of knowledge and skills will be evaluated, as well as the improvement of quality of care based on clinical indicators.

Discussion: The Family Physician is in a privileged situation to increase the performance of the ultrasound in frequent clinical situations and allows a reduction of the attention times. Investigators hope that the results obtained in this study demonstrate the effectiveness of the structured training method (AECAP) and support the generalization of ultrasound in Primary Health Care.

DETAILED DESCRIPTION:
2.1. Design and scope This is a quasi-experimental study, with a before / after design, in which a control group It will be used, with one year of follow-up to evaluate the effectiveness of the training intervention in clinical ultrasound to family doctors. The control group will be composed of family doctors of similar characteristics, who do not participate in the AECAP. The project will be developed with family doctors working in Spanish primary health care centers.

2.2. Study population 20 family doctors who want to participate voluntarily and meet the following inclusion criteria will be included in the study: 1) Physicians should work in a Spanish primary health care center where there is an availability of ultrasound, belonging to the Health Service of Castilla and León (Sacyl) and the Salamanca Health Area. 2.- They must have a list of patients over 800. 3.- Participants must lack prior training in clinical ultrasound. 4.- Participantsmust sign a commitment of assistance and participation in the AECAP. A selection of the control group will be made, with family doctors of similar characteristics, in terms of age, gender, training, work center and number of assigned patients. Participants will be recruited in the first quarter of 2020.

2.3.-Intervention The intervention designed in the AECAP consists of a basic structure and a specific methodology, which will be developed in the teaching classroom of the San Juan Health Center in Salamanca.

Structure: The Material necessary for the realization of the training activity will be: Esaote MyLab ™ Six Echograph (Esaote Spain, Barcelona, Spain); Esaote MyLab ™ Gamma portable ultrasound, a 56-inch high resolution TV with HDMI connection to ultrasound; Fixed computer connected to ultrasound and TV and examination table.

AECAP training methodology: The ultrasound classroom will be biweekly, on the second and fourth Tuesdays of each month, from 6:00 p.m. to 8:30 p.m. At the beginning of the AECAP, the necessary material will be delivered to individually complete the ultrasound training and will be developed with the following structure.

Basic course of clinical ultrasound (abdominal and thyroid) lasting 30 hours, of which 15 hours are theoretical and 15 hours are practical. The course will take place in the first quarter of 2020.

Clinical sessions with patients. At this stage, participants verify the practical usefulness of clinical ultrasound through clinical cases with real patients, who have agreed to participate by signing the informed consent. The sessions will be presented following a structured clinical methodology with a clinical session format with a real patient with the following steps. Before the patient enters the classroom, the clinical case is presented to the participating physicians, then the patient enters to perform the ultrasound with visualization on the classroom screen and written report on the result (Figure 1). All data is incorporated into the "Case Presentation Model. This phase will take place from April to October 2020. The monitor of each session will collect the informed consent of the participating patients.

Final practice: All students must present during the training process, a clinical case in which the use of ultrasound is useful for diagnosis, which will be used to assess the training process. In each clinical case the following variables will be recorded: relevance of ultrasound in the case, agreement of results with clinical data and registration of therapeutic plan and need to perform ultrasound by radiology service or the request for other imaging tests (CT, MRI) ) and endoscopies.

Evaluation of the intervention: Primary and secondary outcomes Primary results: Assessment of knowledge and skills. An initial knowledge evaluation will be carried out, prior to the beginning of the training intervention consisting of 10 single-type test questions: 5 theoretical questions about the basis and use of ultrasound and 5 images to interpret pathologies or ultrasound anatomy. Once the training sessions and practices are started, a continuous evaluation system will be used through which students will be evaluated by teachers / monitors, assessing in a standardized way, theoretical, practical and interpretative aspects. For the final evaluation, on the one hand, a new test of 10 test questions similar to the initial one (5 of theory and 5 of common images) will be carried out. On the other hand, there will be a structured assessment of the presentation of the final clinical case by each student. Finally, the ultrasound examination of 6 patients with common pathologies or normal ultrasound, who have an abdominal or thyroid ultrasound, previously informed by the radiology service, assessing concordance in the description, measures and diagnosis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. -Physicians should work in a Spanish primary health care center with ultrasound,
2. - They must have a list of patients over 800.
3. - They must lack prior training in clinical ultrasound.
4. - They must sign a commitment of assistance and participation in the AECAP

Exclusion Criteria:

1.- No ultrasound availability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of Knowledge by questionaire | 1 year
  A knowledge assessment will be carried out, prior to the start of the training intervention consisting of 10 single-type test questions

SECONDARY OUTCOMES:
Evaluation of outcome in clinical practice. | 1 year
  Diagnostic Delay Times

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research Unit of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Diego-Dominguez F, Torrecilla-Garcia M, Casado-Huerga J, Paule-Sanchez MA, Soria-Lopez CI, Iglesias-Clemente JM, de Dios-Hernandez JM, Diego-Mangas N, Cubillo-Jimenez M, Perez-Escanilla F. Effectiveness of a primary care clinical ultrasound classroom for family physicians as a formative intervention system, a quasi-experimental trial: Study protocol. Medicine (Baltimore). 2020 Jul 2;99(27):e19914. doi: 10.1097/MD.0000000000019914. PMID 32629625